CLINICAL TRIAL: NCT01043666
Title: Phase III Study of YM178: A Randomized, Double-blind, Parallel Group, Placebo and Active Controlled, Multi-center Study in Subjects With Symptoms of Overactive Bladder
Brief Title: A Study of YM178 in Subjects With Symptoms of Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 178-CL-090
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Micturition; YM178; Urinary incontinence; Frequency; Overactive Bladder; Urgency; Urinary urge incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Urinary Incontinence, Urge | interventions — mirabegron; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- YM178 group (Experimental): oral
  Interventions: Drug: YM178
- placebo group (Placebo Comparator): oral
  Interventions: Drug: Placebo
- tolterodine ER group (Experimental): oral
  Interventions: Drug: tolterodine ER

INTERVENTIONS:
Drug: YM178 — oral
  Other Names: mirabegron
  Arms: YM178 group
Drug: Placebo — oral
  Arms: placebo group
Drug: tolterodine ER — oral
  Other Names: Detrusitol SR
  Arms: tolterodine ER group

SUMMARY:
This study is to assess the efficacy and safety of YM178 in patients with symptoms of overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptoms of overactive bladder for at least 12 weeks before the study
* Subjects capable of walking to the lavatory without assistance and measuring the urine volume by him/herself
* Subject with an average frequency of micturition of 8 or more times per 24-hour period
* Subject with an average episode of urgency or urge incontinence of one or more times per 24-hours period
* Subject having provided written informed consent by him/herself

Exclusion Criteria:

* Subject having stress urinary incontinence as a predominant symptom
* Subject with transient symptoms suspected for overactive bladder
* Subject complicated with urinary tract infection, urinary stones, and/or interstitial cystitis or with a historical condition of recurrent urinary tract infection
* Subject complicated with bladder tumor/prostatic tumor or with the historical condition
* Subject confirmed to have a post-void residual volume of >=100ml or with a clinically significant lower urinary tract obstructive disease
* Subject with indwelling catheter or practicing intermittent self-catheterization
* Subject giving radiotherapy influencing urinary tract functions, or thermotherapy for benign prostatic hyperplasia
* Subject giving surgical therapy which may influence urinary tract functions within 24 weeks before the study
* Subject with uncontrolled hypertension (indicated by sitting SBP >=180mmHg or DPB >= 110mmHg)
* Subject with a pulse rate >= 110bpm or <50 bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1126 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2011-09-16 (Actual); Study Completion 2011-09-16 (Actual)

PRIMARY OUTCOMES:
Change in mean number of micturitions per 24 hrs | Within a 12-week treatment period

SECONDARY OUTCOMES:
Change in mean number of urgency episodes per 24 hrs | Within a 12-week treatment period
Change in mean number of urinary incontinence episodes per 24 hrs | Within a 12-week treatment period
Change in mean number of urge incontinence episodes per 24 hrs | Within a 12-week treatment period
Change in mean volume voided per micturition | Within a 12-week treatment period
Change in mean number of nocturia episodes | Within a 12-week treatment period
Safety assessed by vital signs, adverse events laboratory findings, 12-lead electrocardiogram and post-void residual volume | During 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (35):
- China (11):
  - Beijing
  - Dalian
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Hubei
  - Hunan
  - Jiangsu
  - Liaoning
  - Nanjing
  - Shanghai
- India (6):
  - Ahmedabad
  - Gūrgaon
  - Jaipur
  - Lucknow
  - New Delhi
  - Pune
- South Korea (11):
  - Busan
  - Chungcheong Namdo
  - Daegu
  - Daejeon
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Jeollabuk
  - Jeollanam
  - Kyonggi
  - Seoul
- Taiwan (7):
  - Chiayi City
  - Hualien City
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=168